CLINICAL TRIAL: NCT02294396
Title: Postmarketing Study of Mirabegron in Japan: Long-term Add-on Therapy With Antimuscarinics in Patients With Overactive Bladder Treated With Mirabegron
Brief Title: Postmarketing Study to Evaluate add-on Therapy With Anticholinergics in Patients With Overactive Bladder (OAB) on Mirabegron.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 178-CL-112
Record Dates: First submitted 2014-11-10; First posted 2014-11-19 (Estimated); Results first posted 2018-12-24 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Overactive Bladder (OAB)
Keywords: Anticholinergic; Overactive Bladder (OAB); Mirabegron; YM178
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — mirabegron; Solifenacin Succinate; propiverine; imidafenacin; Tolterodine Tartrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Mirabegron + Solifenacin (Experimental): Participants received mirabegron 50 mg and solifenacin 5 mg once daily after breakfast orally for 8 weeks. In the next 44 weeks, participants continued to receive mirabegron 50 mg, but received an increased dose of solifenacin 10 mg, if the treatment was not effective.
  Interventions: Drug: Mirabegron tablet; Drug: Solifenacin tablet
- Mirabegron + Propiverine (Experimental): Participants received mirabegron 50 mg and propiverine 20 mg once daily after breakfast orally for 8 weeks. In the next 44 weeks, participants continued to receive mirabegron 50 mg, but received an increased dose of propiverine 40 mg, if the treatment was not effective.
  Interventions: Drug: Mirabegron tablet; Drug: Propiverine tablet
- Mirabegron + Imidafenacin (Experimental): Participants received mirabegron 50 mg and imidafenacin 0.2 mg once daily after breakfast orally for 8 weeks. In the next 44 weeks, participants continued to receive mirabegron 50 mg, but received an increased dose of imidafenacin 0.4 mg, if the treatment was not effective.
  Interventions: Drug: Mirabegron tablet; Drug: Imidafenacin tablet
- Mirabegron + Tolterodine (Experimental): Participants received mirabegron 50 mg and tolterodine 4 mg once daily after breakfast orally for 52 weeks.
  Interventions: Drug: Mirabegron tablet; Drug: Tolterodine capsule

INTERVENTIONS:
Drug: Mirabegron tablet — orally administered at a dose of 1 tablet once daily after breakfast
  Other Names: YM178
Drug: Solifenacin tablet — orally administered at a dose of 1 tablet once daily after breakfast (could be increased to 2 tablets)
  Arms: Mirabegron + Solifenacin
Drug: Propiverine tablet — orally administered at a dose of 1 tablet once daily after breakfast (could be increased to 1 tablet twice daily after breakfast and after dinner)
  Arms: Mirabegron + Propiverine
Drug: Imidafenacin tablet — orally administered at a dose of 1 tablet (0.1 mg tablet) twice daily after breakfast and after dinner (could be increased to 2 tablets twice daily after breakfast and after dinner)
  Arms: Mirabegron + Imidafenacin
Drug: Tolterodine capsule — orally administered at a dose of 1 capsule once daily after breakfast (could not be increased)
  Arms: Mirabegron + Tolterodine

SUMMARY:
The objective of the study was to evaluate the safety and efficacy of add-on therapy with anticholinergics in patients with OAB on mirabegron.

DETAILED DESCRIPTION:
This was a multicenter, open-label study to evaluate the safety and efficacy of add-on therapy with antimuscarinics in patients with OAB treated with mirabegron.

The total duration of the study period was 54 weeks in total, comprising a 2-week screening period and a 52-week treatment period. Patients who met the eligibility criteria for provisional enrollment received orally the study drug for the screening period (mirabegron 50 mg) once daily after breakfast for 2 weeks. Patients who met the eligibility criteria after the screening period were randomized to solifenacin 5 mg, propiverine 20 mg, imidafenacin 0.2 mg or tolterodine 4 mg in a 1:1:1:1 ratio, and received orally mirabegron 50 mg and antimuscarinics for 52 weeks. At week 8 visit, the dose of all antimuscarinics except for tolterodine could be increased by 2-fold (solifenacin 10 mg, propiverine 40 mg or imidafenacin 0.4 mg) if a patient met the following criteria: (1) had no response to the study drugs; (2) was considered by the investigator to have no safety concerns; and (3) agreed to increase the dose. However, in the event of AEs after the dose was increased, it could be reduced to the level before the increase. A dose increase for a second time after dose reduction was not permitted.

ELIGIBILITY:
Inclusion Criteria:

* Female: OAB outpatient who had been postmenopausal for at least 1 year
* Male: OAB outpatient who had no wish to have children in the future
* Patient had been under treatment with mirabegron at a stable dose of 50 mg once daily for at least 6 weeks before the start of the screening period
* Patient capable of walking to the bathroom without assistance
* Patient had a total Overactive Bladder Symptom Score (OABSS) of ≥3 points and a Question 3 score of ≥2 points

Exclusion Criteria:

* Patient had an established diagnosis of stress urinary incontinence (patient had no symptom other than stress urinary incontinence)
* Patient had urinary tract infection (cystitis, prostatitis, etc.), urinary calculus (ureteric calculus, urethral calculus, bladder calculus, etc.), interstitial cystitis, or a history of recurrent urinary tract infection (at least 3 episodes within 24 weeks before the start of the screening period)
* Patient had a residual urine volume of ≥100 mL at week -2 visit or patient with benign prostatic hyperplasia or lower urinary tract obstruction
* Patient had uncontrolled hypertension (sitting systolic blood pressure ≥180 mmHg or diastolic blood pressure ≥110 mmHg at week -2 visit)
* Patient had a pulse rate of ≥110 bpm or <50 bpm at week -2 visit
* Patient had a contraindication to antimuscarinics (urinary retention; obstruction in thepylorus, duodenum, or intestine; paralytic ileus; gastric/intestinal atony; myasthenia gravis; and decreased gastrointestinal motility/tone, etc.)
* Patient had glaucoma, ulcerative colitis, hyperthyroidism, dementia, cognitive dysfunction, parkinsonism symptoms, or clinically significant cerebrovascular disorder
* Patient had serious heart disease (myocardial infarction, cardiac failure, uncontrolled angina pectoris, serious arrhythmia, use of pacemaker, etc.), liver disease, kidney disease, immunological disease, lung disease, etc. or patient had a history of malignant tumor (except for malignant tumor that had not been treated for at least 5 years before the start of the screening period with no risk of recurrence)
* Patient had drug hypersensitivity to β-agonists or anticholinergics
* Patient was under treatment with flecainide acetate or propafenone hydrochloride
* Patient had long QT syndrome, patient was vulnerable to arrhythmia such as bradycardia or acute myocardial ischemia, patient had hypokalemia, and patient had ischemic heart disease such as angina pectoris
* Patient had used any prohibited concomitant medication within 4 weeks before the start of the screening period
* Patient was under catheterization or intermittent self-catheterization or patient had pelvic organ prolapse that affected the urinary tract function
* Patient had received radiotherapy that affected the urinary tract function
* Patient had received surgical therapy that may have affected the urinary tract function within 24 weeks before the start of the screening period
* Patient had received nonpharmacological therapy for OAB such as electric stimulation therapy (interferential low frequency therapy, magnetic stimulation therapy, etc.), biofeedback therapy, bladder training, or pelvic floor muscle exercise within 2 weeks before the start of the screening period
* Patient had or had a history of mood disorder, neurotic disorder, and schizophrenia

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 649 (Actual)
Dates: Start 2014-10-28 (Actual); Primary Completion 2016-09-07 (Actual); Study Completion 2016-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (7):
- Japan (7):
  - Chugoku
  - Chūbu
  - Hokkaido
  - Kansai
  - Kantou
  - Kyushu
  - Tōhoku

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/study.aspx?ID=224

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with overactive bladder (OAB) were enrolled in 60 sites in Japan.
Pre-assignment Details: Prior to randomization, participants received 50 mg mirabegron orally once daily after breakfast for 2 weeks during a screening period.
Period: Overall Study
Arm/Group | Mirabegron + Solifenacin | Mirabegron + Propiverine | Mirabegron + Imidafenacin | Mirabegron + Tolterodine
Started | 167 | 161 | 161 | 160
Completed | 127 | 128 | 126 | 123
Not Completed | 40 | 33 | 35 | 37
Not completed — Adverse Event | 26 | 25 | 21 | 24
Not completed — Electrocardiogram adviser's judgment | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 8 | 6 | 6 | 8
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1
Not completed — Protocol Deviation | 3 | 2 | 2 | 1
Not completed — Miscellaneous | 2 | 0 | 5 | 2

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAF). The SAF consisted of participants who received at least 1 dose of the study drug for the treatment period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Mirabegron + Solifenacin | Mirabegron + Propiverine | Mirabegron + Imidafenacin | Mirabegron + Tolterodine | Total
Number analyzed (Participants) | 166 | 161 | 161 | 159 | 647
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (9.4) | 64.0 (9.3) | 65.7 (8.7) | 65.7 (10.0) | 65.0 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 146 | 144 | 146 | 134 | 570
  Male | 20 | 17 | 15 | 25 | 77
Overactive Bladder Symptom Score (OABSS) [Mean (Standard Deviation); unit: Units on a Scale] — The OABSS questionnaire was a questionnaire completed by participants with 4 questions regarding their OAB symptoms. For each participant, the OABSS total score was calculated from the sum total of the score of each question. The total score ranges from 0 to 15 with higher score indicating more symptoms. The OABSS data obtained at week 0 were used as baseline. Population: Full Analysis Set (FAS). The FAS consisted of participants who received at least 1 dose of the study drugs for the treatment period and who provided evaluable efficacy data for at least 1 variable before and after the start of the treatment period. Participants with available data are included in the analysis.
  Units on a Scale | 7.4 (2.6) | 7.7 (2.5) | 7.8 (2.3) | 7.7 (2.3) | 7.6 (2.4)
Overactive Bladder questionnaire Short Form (OAB-q SF) Score: Symptom Severity [Mean (Standard Deviation); unit: Units on a Scale] — The OAB-q SF questionnaire was a questionnaire completed by participants composed of 2 sections: Severity Symptom and the Health-related Quality of Life (HRQL). The Severity Symptom section included 6 questions. For each participant, the symptom severity score was derived as a sum of scores for Questions 1 to 6. The total score ranges from 6 to 36 with higher symptom severity score indicating greater symptom bother. OAB-q SF data obtained at week 0 visit were used as baseline. Population: FAS participants with available data are included in the analysis.
  Units on a Scale | 32.81 (20.78) | 32.36 (21.23) | 32.92 (19.45) | 34.23 (22.60) | 33.08 (21.00)
OAB-q SF Score: Total Health-Related Quality of Life (HRQOL) [Mean (Standard Deviation); unit: Units on a Scale] — The OAB-q SF questionnaire was a questionnaire completed by participants composed of 2 sections: Severity Symptom and the HRQL. The HRQL section included 13 questions. For each participant, the total HRQL score was derived as a sum of scores for Questions 7 to 19. The total score ranges from 13 to 78 with higher total HRQL score indicating greater HRQL. OAB-q SF data obtained at week 0 visit were used as baseline. Population: FAS participants with available data are included in the analysis.
  Units on a Scale | 75.16 (17.65) | 77.36 (16.11) | 74.85 (18.50) | 75.37 (19.33) | 75.68 (17.91)
Mean Number of Micturitions per 24 Hours [Mean (Standard Deviation); unit: micturitions] — The mean number of micturitions per 24 hours was calculated by taking the sum of all marked episodes in the patient diary where the variable "urinated" was indicated, divided by the number of days on which episodes were recorded. Population: FAS participants with available data are included in the analysis.
  micturitions | 10.06 (2.59) | 10.37 (2.65) | 10.13 (2.92) | 10.20 (2.62) | 10.19 (2.69)
Mean Number of Urgency Episodes per 24 Hours [Mean (Standard Deviation); unit: urgency episodes] — An urgency episode was defined as a complaint of a sudden, compelling desire to pass urine, which is difficult to defer. The mean number of urgency episodes per 24 hours was calculated by taking the sum of all marked episodes in the patient diary where the variable "urgency" was indicated, divided by the number of days on which episodes were recorded. Only participants who had an urgency episode at baseline was included in the analysis. Population: FAS participants with available data are included in the analysis.
  urgency episodes
    number analyzed (Participants) | 153 | 148 | 150 | 148 | 599
    (all) | 3.26 (2.46) | 3.12 (2.67) | 3.27 (2.20) | 3.15 (2.54) | 3.20 (2.47)
Mean Number of Incontinence Episodes per 24 Hours [Mean (Standard Deviation); unit: incontinence episodes] — An incontinence episode was defined as the complaint of any involuntary leakage of urine. The mean number of incontinence episodes per 24 hours was calculated by taking the sum of all marked episodes in the patient diary where the variable "urinary incontinence'" was indicated, divided by the number of days on which episodes were recorded. Only participants who had an incontinence episode at baseline was included in the analysis. Population: FAS participants with available data are included in the analysis.
  incontinence episodes
    number analyzed (Participants) | 91 | 95 | 103 | 96 | 385
    (all) | 1.62 (1.62) | 1.59 (1.83) | 1.47 (1.35) | 1.55 (1.76) | 1.56 (1.64)
Mean Number of Urge Incontinence Episodes per 24 Hours [Mean (Standard Deviation); unit: urge incontinence episodes] — An urge incontinence episode was defined as any episode when both urgency and incontinence occurred concurrently. The mean number of incontinence episodes per 24 hours was calculated by taking the sum of all marked episodes in the patient diary where the variable "urgency" and "urinary incontinence'" were indicated, divided by the number of days on which episodes were recorded. Only participants who had an urge incontinence episode at baseline was included in the analysis. Population: FAS participants with available data are included in the analysis.
  urge incontinence episodes
    number analyzed (Participants) | 80 | 82 | 86 | 85 | 333
    (all) | 1.55 (1.47) | 1.39 (1.45) | 1.30 (1.16) | 1.31 (1.62) | 1.38 (1.43)
Mean Volume Voided per Micturition [Mean (Standard Deviation); unit: mL] — The mean volume per micturition was calculated by taking the sum of the urinary volumes where the volume voided was > 0 and where "urinary incontinence" was not indicated in the patient diary, divided by the number of micturitions where the volume voided was > 0 and where "urinary incontinence" was not indicated. Only participants who had volume voided was > 0 at baseline was included in the analysis. Population: FAS participants with available data are included in the analysis.
  mL | 166.600 (50.404) | 170.064 (63.781) | 169.309 (50.324) | 167.542 (54.320) | 168.368 (54.839)
Mean Number of Nocturia Episodes per Night [Mean (Standard Deviation); unit: nocturia episodes] — A nocturia episode was defined as waking at night 1 or more times to void. Night time was defined as the period between bedtime and the wake-up time the following day (micturitions at the same time as the wake-up time were excluded). The mean number of nocturia episodes per night was calculated by taking the sum of nocturia episodes in the patient diary where the variable "urinated" was indicated during the night time, divided by the number of nights. Only participants who had a nocturia episode at baseline was included in the analysis. Population: FAS participants with available data are included in the analysis.
  nocturia episodes
    number analyzed (Participants) | 142 | 133 | 141 | 132 | 548
    (all) | 1.50 (0.96) | 1.68 (1.08) | 1.61 (1.29) | 1.67 (1.04) | 1.61 (1.10)
Postvoid Residual (PVR) Volume [Mean (Standard Deviation); unit: mL] — Measurement of PVR volume was made using either ultrasonography or urethral catheterization, provided that the same method was used for the same participant throughout the study.
  mL | 11.02 (15.43) | 10.43 (17.07) | 9.74 (14.35) | 9.10 (14.41) | 10.08 (15.34)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: TEAEs were defined as AEs observed after the first administration of the study drugs for the treatment period. The investigator assessed the severity of AEs, including abnormal clinical laboratory values, electrocardiogram (ECG), vital signs, as follows: Mild: No disruption of normal daily activities; Moderate: Affected normal daily activities; Severe: Inability to perform daily activities. A drug-related TEAE was a TEAE with at least a possible relationship to the study drug as assessed by the investigator.
Time Frame: From first dose of study drug up to week 52
Population: SAF
Measure: Count of Participants; unit: Participants
Arm/Group | Mirabegron + Solifenacin | Mirabegron + Propiverine | Mirabegron + Imidafenacin | Mirabegron + Tolterodine
Number analyzed (Participants) | 166 | 161 | 161 | 159
Participants
  Any TEAEs | 131 | 135 | 133 | 120
  Mild | 113 | 122 | 116 | 104
  Moderate | 15 | 13 | 15 | 12
  Severe | 3 | 0 | 2 | 4
  Drug-related TEAEs | 76 | 81 | 72 | 74
  TEAEs leading to death | 0 | 0 | 0 | 1
  Drug-related TEAEs leading to death | 0 | 0 | 0 | 0
  Serious TEAEs | 10 | 4 | 5 | 9
  Drug-related serious TEAEs | 0 | 1 | 0 | 1
  TEAEs leading to withdrawal of treatment | 23 | 19 | 16 | 18
  Drug-related TEAEs leading to withdrawal of treat. | 12 | 17 | 10 | 8

2. Secondary Outcome: Change From Baseline in Overactive Bladder Symptom Score (OABSS) Total Score
Description: The OABSS questionnaire was a questionnaire completed by participants with 4 questions regarding their OAB symptoms. For each participant, the OABSS total score was calculated from the sum total of the score of each question. The total score ranges from 0 to 15 with higher score indicating more symptoms. The OABSS data obtained at week 0 were used as baseline.
Time Frame: Baseline and week 4, 8, 12, 16, 28 and 52
Population: FAS participants with available data at each time point are included in the analysis. A last visit analysis (at the end of treatment) was performed to ensure all participants with postbaseline data were included in the analyses. Last observation carried forward (LOCF) imputation was used for the end of treatment analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mirabegron + Solifenacin | Mirabegron + Propiverine | Mirabegron + Imidafenacin | Mirabegron + Tolterodine
Number analyzed (Participants) | 166 | 161 | 161 | 159
units on a scale
  Week 4: number analyzed (Participants) | 162 | 157 | 158 | 157
  Week 4 | -2.9 (2.5) | -3.1 (2.5) | -2.4 (2.3) | -3.0 (2.5)
  Week 8: number analyzed (Participants) | 155 | 148 | 155 | 147
  Week 8 | -3.5 (2.5) | -3.7 (2.5) | -3.1 (2.3) | -3.5 (2.6)
  Week 12: number analyzed (Participants) | 144 | 146 | 145 | 142
  Week 12 | -4.0 (2.6) | -4.2 (2.8) | -3.4 (2.2) | -4.0 (2.6)
  Week 16: number analyzed (Participants) | 138 | 140 | 144 | 137
  Week 16 | -4.1 (2.7) | -4.4 (2.7) | -3.8 (2.3) | -4.4 (2.6)
  Week 28: number analyzed (Participants) | 133 | 133 | 140 | 133
  Week 28 | -4.0 (2.6) | -4.4 (2.9) | -3.9 (2.8) | -4.3 (2.9)
  Week 52: number analyzed (Participants) | 127 | 128 | 125 | 123
  Week 52 | -4.0 (2.7) | -4.1 (2.5) | -4.1 (2.6) | -4.3 (2.9)
  End of treatment: number analyzed (Participants) | 164 | 160 | 161 | 159
  End of treatment | -3.9 (2.7) | -4.1 (2.6) | -3.9 (2.6) | -4.2 (2.8)

3. Secondary Outcome: Number of Participants Who Achieved Normalization for OABSS Total Score
Description: Normalization for OABSS Total Score was defined as OABSS total score ≤ 2 or OABSS Question 3 score ≤ 1.
Time Frame: Week 52 (end of treatment)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Mirabegron + Solifenacin | Mirabegron + Propiverine | Mirabegron + Imidafenacin | Mirabegron + Tolterodine
Number analyzed (Participants) | 164 | 160 | 161 | 159
Participants | 98 | 101 | 91 | 96

4. Secondary Outcome: Change From Baseline in Overactive Bladder Questionnaire Short Form (OAB-q SF) Symptom Severity Score
Description: The OAB-q SF questionnaire was a questionnaire completed by participants composed of 2 sections: Symptom Severity and the Health-related Quality of Life (HRQL). The Symptom Severity section included 6 questions. For each participant, the symptom severity score was derived as a sum of scores for Questions 1 to 6. The total score ranges from 6 to 36 with higher symptom severity score indicating greater symptom bother. OAB-q SF data obtained at week 0 visit were used as baseline.
Time Frame: Baseline and week 12, 28 and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mirabegron + Solifenacin | Mirabegron + Propiverine | Mirabegron + Imidafenacin | Mirabegron + Tolterodine
Number analyzed (Participants) | 166 | 161 | 161 | 159
units on a scale
  Week 12: number analyzed (Participants) | 144 | 146 | 145 | 142
  Week 12 | -18.59 (15.89) | -20.2 (19.40) | -17.15 (17.37) | -21.22 (20.42)
  Week 28: number analyzed (Participants) | 133 | 133 | 140 | 133
  Week 28 | -21.38 (18.15) | -21.40 (19.18) | -20.40 (19.23) | -21.95 (20.95)
  Week 52: number analyzed (Participants) | 127 | 128 | 125 | 123
  Week 52 | -20.55 (18.29) | -20.68 (19.33) | -20.51 (18.28) | -22.49 (21.23)
  End of treatment: number analyzed (Participants) | 160 | 159 | 159 | 154
  End of treatment | -18.92 (18.42) | -18.99 (19.14) | -18.89 (18.11) | -21.28 (20.99)

5. Secondary Outcome: Change From Baseline in OAB-q SF Total HRQL Score
Description: The OAB-q SF questionnaire was a questionnaire completed by participants composed of 2 sections: Severity Symptom and the HRQL. The HRQL section included 13 questions. For each participant, the total HRQL score was derived as a sum of scores for Questions 7 to 19. The total score ranges from 13 to 78 with higher total HRQL score indicating greater HRQL. OAB-q SF data obtained at week 0 visit were used as baseline.
Time Frame: Baseline and week 12, 28 and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mirabegron + Solifenacin | Mirabegron + Propiverine | Mirabegron + Imidafenacin | Mirabegron + Tolterodine
Number analyzed (Participants) | 166 | 161 | 161 | 159
units on a scale
  Week 12: number analyzed (Participants) | 144 | 146 | 145 | 142
  Week 12 | 12.07 (13.37) | 11.35 (13.15) | 11.06 (15.72) | 12.05 (16.00)
  Week 28: number analyzed (Participants) | 133 | 133 | 140 | 133
  Week 28 | 15.15 (14.63) | 13.05 (14.00) | 14.88 (17.16) | 12.94 (15.55)
  Week 52: number analyzed (Participants) | 127 | 128 | 125 | 123
  Week 52 | 15.99 (14.63) | 13.89 (14.04) | 14.67 (16.88) | 15.06 (16.40)
  End of treatment: number analyzed (Participants) | 160 | 159 | 159 | 154
  End of treatment | 14.38 (14.98) | 12.46 (13.89) | 13.99 (16.72) | 14.36 (17.51)

6. Secondary Outcome: Change From Baseline in the Mean Number of Micturitions Per 24 Hours
Description: Participants completed the patient diary (paper document) for 3 days immediately before each visit. The mean number of micturitions per 24 hours was calculated by taking the sum of all marked episodes in the patient diary where the variable "urinated" was indicated, divided by the number of days on which episodes were recorded.
Time Frame: Baseline and week 4, 8, 12, 16, 28, 40, 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: micturitions
Arm/Group | Mirabegron + Solifenacin | Mirabegron + Propiverine | Mirabegron + Imidafenacin | Mirabegron + Tolterodine
Number analyzed (Participants) | 166 | 161 | 161 | 159
micturitions
  Week 4: number analyzed (Participants) | 158 | 155 | 157 | 156
  Week 4 | -1.57 (1.52) | -1.44 (1.70) | -1.23 (1.80) | -1.51 (1.84)
  Week 8: number analyzed (Participants) | 154 | 148 | 153 | 146
  Week 8 | -1.85 (1.69) | -1.89 (1.87) | -1.62 (1.95) | -1.72 (1.87)
  Week 12: number analyzed (Participants) | 142 | 146 | 145 | 142
  Week 12 | -2.04 (1.74) | -1.90 (1.96) | -1.74 (1.90) | -2.18 (2.10)
  Week 16: number analyzed (Participants) | 137 | 138 | 144 | 137
  Week 16 | -2.33 (1.74) | -2.21 (2.03) | -1.86 (2.00) | -2.20 (2.07)
  Week 28: number analyzed (Participants) | 132 | 134 | 139 | 132
  Week 28 | -2.29 (2.05) | -2.10 (2.16) | -1.97 (2.39) | 2.33 (2.09)
  Week 40: number analyzed (Participants) | 128 | 130 | 130 | 126
  Week 40 | -2.12 (2.01) | -1.97 (2.17) | -1.80 (2.14) | -1.92 (1.90)
  Week 52: number analyzed (Participants) | 127 | 128 | 125 | 123
  Week 52 | -2.29 (2.01) | -2.08 (2.11) | -1.82 (2.16) | -1.80 (2.10)
  End of treatment: number analyzed (Participants) | 159 | 155 | 157 | 156
  End of treatment | -2.18 (1.96) | -1.89 (2.08) | -1.75 (2.09) | -1.91 (2.22)

7. Secondary Outcome: Number for Participants Who Achieved Normalization of the Mean Number of Micturitions Per 24 Hours
Description: Normalization for the mean number of micturitions per 24 hours was defined as < 8 micturitions per 24 hours.
Time Frame: Week 52 (end of treatment)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Mirabegron + Solifenacin | Mirabegron + Propiverine | Mirabegron + Imidafenacin | Mirabegron + Tolterodine
Number analyzed (Participants) | 159 | 155 | 157 | 156
Participants | 60 | 47 | 47 | 51

8. Secondary Outcome: Change From Baseline in the Mean Number of Urgency Episodes Per 24 Hours
Description: Participants completed the patient diary (paper document) for 3 days immediately before each visit. An urgency episode was defined as a complaint of a sudden, compelling desire to pass urine, which is difficult to defer. The mean number of urgency episodes per 24 hours was calculated by taking the sum of all marked episodes in the patient diary where the variable "urgency" was indicated, divided by the number of days on which episodes were recorded. Only participants who had an urgency episode at baseline was included in the analysis.
Time Frame: Baseline and week 4, 8, 12, 16, 28, 40, 52
Population: FAS participants with available data at each time point are included in the analysis.A last visit analysis (at the end of treatment) was performed to ensure all participants with postbaseline data were included in the analyses. Last observation carried forward (LOCF) imputation was used for the end of treatment analysis.
Measure: Mean (Standard Deviation); unit: urgency episodes
Arm/Group | Mirabegron + Solifenacin | Mirabegron + Propiverine | Mirabegron + Imidafenacin | Mirabegron + Tolterodine
Number analyzed (Participants) | 153 | 148 | 150 | 148
urgency episodes
  Week 4: number analyzed (Participants) | 146 | 143 | 149 | 146
  Week 4 | -1.53 (1.99) | -1.63 (2.20) | -1.23 (1.62) | -1.49 (2.16)
  Week 8: number analyzed (Participants) | 142 | 139 | 145 | 137
  Week 8 | -1.78 (2.13) | -1.90 (2.20) | -1.50 (1.65) | -1.89 (2.24)
  Week 12: number analyzed (Participants) | 132 | 137 | 137 | 132
  Week 12 | -2.06 (2.20) | -2.18 (2.39) | -1.88 (1.78) | -2.10 (2.23)
  Week 16: number analyzed (Participants) | 127 | 129 | 136 | 129
  Week 16 | -2.30 (2.22) | -2.36 (2.56) | -2.01 (1.89) | -2.26 (2.30)
  Week 28: number analyzed (Participants) | 122 | 127 | 132 | 124
  Week 28 | -2.28 (2.25) | -2.26 (2.76) | -2.18 (2.10) | -2.28 (2.39)
  Week 40: number analyzed (Participants) | 118 | 123 | 125 | 119
  Week 40 | -2.14 (2.33) | -2.27 (2.64) | -2.14 (2.17) | -2.19 (2.42)
  Week 52: number analyzed (Participants) | 117 | 121 | 119 | 117
  Week 52 | -2.04 (2.69) | -2.33 (2.54) | -2.15 (2.28) | -2.26 (2.31)
  End of treatment: number analyzed (Participants) | 147 | 143 | 149 | 146
  End of treatment | -2.03 (2.55) | -2.24 (2.41) | -2.04 (2.19) | -2.07 (2.23)

9. Secondary Outcome: Number for Participants Who Achieved Normalization of the Mean Number of Urgency Episodes Per 24 Hours
Description: Normalization for the mean number of urgency episodes per 24 hours was defined as no urgency episode per 24 hours.
Time Frame: Week 52 (end of treatment)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Mirabegron + Solifenacin | Mirabegron + Propiverine | Mirabegron + Imidafenacin | Mirabegron + Tolterodine
Number analyzed (Participants) | 147 | 143 | 149 | 146
Participants | 70 | 77 | 64 | 76

10. Secondary Outcome: Change From Baseline in the Mean Number of Incontinence Episodes Per 24 Hours
Description: Participants completed the patient diary (paper document) for 3 days immediately before each visit. An incontinence episode was defined as the complaint of any involuntary leakage of urine. The mean number of incontinence episodes per 24 hours was calculated by taking the sum of all marked episodes in the patient diary where the variable "urinary incontinence'" was indicated, divided by the number of days on which episodes were recorded. Only participants who had an incontinence episode at baseline was included in the analysis.
Time Frame: Baseline and week 4, 8, 12, 16, 28, 40, 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: incontinence episodes
Arm/Group | Mirabegron + Solifenacin | Mirabegron + Propiverine | Mirabegron + Imidafenacin | Mirabegron + Tolterodine
Number analyzed (Participants) | 91 | 94 | 102 | 95
incontinence episodes
  Week 4: number analyzed (Participants) | 87 | 92 | 101 | 93
  Week 4 | -1.13 (1.40) | -1.06 (1.50) | -0.81 (0.95) | -1.09 (1.66)
  Week 8: number analyzed (Participants) | 86 | 88 | 97 | 89
  Week 8 | -1.16 (1.44) | -1.21 (1.50) | -0.74 (1.13) | -1.21 (1.70)
  Week 12: number analyzed (Participants) | 82 | 86 | 92 | 85
  Week 12 | -1.27 (1.44) | -1.34 (1.66) | -0.86 (1.06) | -1.23 (1.58)
  Week 16: number analyzed (Participants) | 79 | 81 | 92 | 82
  Week 16 | -1.23 (1.42) | -1.32 (1.74) | -0.97 (1.02) | -1.33 (1.72)
  Week 28: number analyzed (Participants) | 76 | 77 | 90 | 81
  Week 28 | -1.31 (1.53) | -1.28 (1.82) | -0.99 (1.21) | -1.28 (1.63)
  Week 40: number analyzed (Participants) | 73 | 75 | 83 | 78
  Week 40 | -1.23 (1.53) | -1.28 (1.56) | -0.96 (0.99) | -1.07 (1.52)
  Week 52: number analyzed (Participants) | 72 | 73 | 84 | 76
  Week 52 | -1.31 (1.49) | -1.29 (1.71) | -1.02 (1.08) | -1.18 (1.64)
  End of treatment: number analyzed (Participants) | 87 | 92 | 101 | 93
  End of treatment | -1.25 (1.48) | -1.18 (1.59) | -1.03 (1.08) | -1.15 (1.52)

11. Secondary Outcome: Number for Participants Who Achieved Normalization of the Mean Number of Incontinence Episodes Per 24 Hours
Description: Normalization for the mean number of incontinence episodes per 24 hours was defined as no incontinence episode per 24 hours.
Time Frame: Week 52 (end of treatment)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Mirabegron + Solifenacin | Mirabegron + Propiverine | Mirabegron + Imidafenacin | Mirabegron + Tolterodine
Number analyzed (Participants) | 87 | 92 | 101 | 93
Participants | 61 | 61 | 69 | 71

12. Secondary Outcome: Change From Baseline in the Mean Number of Urge Incontinence Episodes Per 24 Hours
Description: Participants completed the patient diary (paper document) for 3 days immediately before each visit. An urge incontinence episode was defined as any episode when both urgency and incontinence occurred concurrently. The mean number of incontinence episodes per 24 hours was calculated by taking the sum of all marked episodes in the patient diary where the variable "urgency" and "urinary incontinence'" were indicated, divided by the number of days on which episodes were recorded. Only participants who had an urge incontinence episode at baseline was included in the analysis.
Time Frame: Baseline and week 4, 8, 12, 16, 28, 40, 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: urge incontinence episodes
Arm/Group | Mirabegron + Solifenacin | Mirabegron + Propiverine | Mirabegron + Imidafenacin | Mirabegron + Tolterodine
Number analyzed (Participants) | 80 | 82 | 85 | 84
urge incontinence episodes
  Week 4: number analyzed (Participants) | 76 | 80 | 85 | 82
  Week 4 | -1.13 (1.24) | -1.00 (1.32) | -0.72 (0.64) | -0.96 (1.63)
  Week 8: number analyzed (Participants) | 75 | 78 | 81 | 79
  Week 8 | -1.15 (1.31) | -1.14 (1.23) | -0.71 (0.96) | -1.05 (1.64)
  Week 12: number analyzed (Participants) | 71 | 76 | 77 | 75
  Week 12 | -1.20 (1.27) | -1.25 (1.39) | -0.79 (0.88) | -1.13 (1.60)
  Week 16: number analyzed (Participants) | 68 | 71 | 77 | 72
  Week 16 | -1.17 (1.24) | -1.22 (1.47) | -0.87 (0.86) | -1.22 (1.64)
  Week 28: number analyzed (Participants) | 65 | 69 | 75 | 71
  Week 28 | -1.26 (1.34) | -1.10 (1.49) | -0.85 (1.15) | -1.18 (1.63)
  Week 40: number analyzed (Participants) | 62 | 67 | 69 | 70
  Week 40 | -1.19 (1.36) | -1.14 (1.28) | -0.91 (0.96) | -1.07 (1.65)
  Week 52: number analyzed (Participants) | 61 | 66 | 69 | 68
  Week 52 | -1.23 (1.32) | -1.14 (1.37) | -0.93 (0.97) | -1.15 (1.68)
  End of treatment: number analyzed (Participants) | 76 | 80 | 85 | 82
  End of treatment | -1.20 (1.32) | -1.12 (1.33) | -0.91 (0.93) | -1.05 (1.59)

13. Secondary Outcome: Change From Baseline in the Mean Volume Voided Per Micturition
Description: Participants completed the patient diary (paper document) for 3 days immediately before each visit. The mean volume per micturition was calculated by taking the sum of the urinary volumes where the volume voided was > 0 and where "urinary incontinence" was not indicated in the patient diary, divided by the number of micturitions where the volume voided was > 0 and where "urinary incontinence" was not indicated. Only participants who had volume voided was > 0 at baseline was included in the analysis.
Time Frame: Baseline and week 4, 8, 12, 16, 28, 40, 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Mirabegron + Solifenacin | Mirabegron + Propiverine | Mirabegron + Imidafenacin | Mirabegron + Tolterodine
Number analyzed (Participants) | 166 | 161 | 161 | 159
mL
  Week 4: number analyzed (Participants) | 158 | 155 | 157 | 155
  Week 4 | 30.677 (37.450) | 30.111 (39.034) | 20.062 (30.816) | 32.854 (41.598)
  Week 8: number analyzed (Participants) | 154 | 148 | 153 | 146
  Week 8 | 38.328 (41.753) | 38.614 (43.030) | 23.820 (35.972) | 35.351 (35.449)
  Week 12: number analyzed (Participants) | 142 | 146 | 145 | 142
  Week 12 | 39.452 (43.802) | 41.433 (45.910) | 27.072 (41.636) | 36.598 (46.230)
  Week 16: number analyzed (Participants) | 137 | 138 | 144 | 137
  Week 16 | 39.952 (46.871) | 40.661 (48.257) | 24.489 (41.184) | 37.786 (44.837)
  Week 28: number analyzed (Participants) | 132 | 134 | 139 | 132
  Week 28 | 36.025 (50.761) | 41.887 (48.797) | 29.873 (48.976) | 34.823 (42.451)
  Week 40: number analyzed (Participants) | 128 | 130 | 130 | 126
  Week 40 | 43.578 (51.692) | 43.102 (52.130) | 29.826 (44.442) | 41.378 (43.053)
  Week 52: number analyzed (Participants) | 127 | 128 | 125 | 123
  Week 52 | 41.744 (47.045) | 40.599 (45.607) | 36.653 (46.041) | 40.548 (48.033)
  End of treatment: number analyzed (Participants) | 159 | 155 | 157 | 156
  End of treatment | 40.004 (45.095) | 38.691 (46.429) | 32.854 (44.481) | 40.683 (46.566)

14. Secondary Outcome: Change From Baseline in the Mean Number of Nocturia Episodes Per Night
Description: Participants completed the patient diary (paper document) for 3 days immediately before each visit. A nocturia episode was defined as waking at night 1 or more times to void. Night time was defined as the period between bedtime and the wake-up time the following day (micturitions at the same time as the wake-up time were excluded). The mean number of nocturia episodes per night was calculated by taking the sum of nocturia episodes in the patient diary where the variable "urinated" was indicated during the night time, divided by the number of nights. Only participants who had a nocturia episode at baseline was included in the analysis.
Time Frame: Baseline and week 4, 8, 12, 16, 28, 40, 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nocturia episodes
Arm/Group | Mirabegron + Solifenacin | Mirabegron + Propiverine | Mirabegron + Imidafenacin | Mirabegron + Tolterodine
Number analyzed (Participants) | 144 | 137 | 143 | 134
nocturia episodes
  Week 4: number analyzed (Participants) | 136 | 131 | 139 | 130
  Week 4 | -0.33 (0.83) | -0.29 (0.73) | -0.32 (1.00) | -0.49 (0.83)
  Week 8: number analyzed (Participants) | 132 | 124 | 135 | 121
  Week 8 | -0.42 (0.82) | -0.37 (0.80) | -0.42 (0.92) | -0.44 (0.85)
  Week 12: number analyzed (Participants) | 121 | 122 | 128 | 116
  Week 12 | -0.45 (0.96) | -0.28 (0.93) | -0.45 (0.99) | -0.47 (0.81)
  Week 16: number analyzed (Participants) | 117 | 117 | 127 | 112
  Week 16 | -0.49 (0.86) | -0.37 (0.92) | -0.54 (0.99) | -0.50 (0.94)
  Week 28: number analyzed (Participants) | 112 | 113 | 121 | 109
  Week 28 | -0.42 (1.00) | -0.39 (0.93) | -0.48 (0.97) | -0.54 (0.81)
  Week 40: number analyzed (Participants) | 108 | 109 | 114 | 103
  Week 40 | -0.53 (0.93) | -0.45 (0.83) | -0.39 (0.94) | -0.54 (0.82)
  Week 52: number analyzed (Participants) | 107 | 107 | 110 | 100
  Week 52 | -0.55 (0.91) | -0.44 (0.86) | -0.53 (0.95) | -0.50 (0.94)
  End of treatment: number analyzed (Participants) | 137 | 131 | 139 | 130
  End of treatment | -0.47 (0.91) | -0.38 (0.88) | -0.48 (0.93) | -0.48 (0.88)

15. Secondary Outcome: Number of Participants Who Achieved Normalization of the Mean Number of Nocturia Episodes Per 24 Hours
Description: Normalization for the mean number of nocturia episodes per 24 hours was defined as no nocturia episode per 24 hours.
Time Frame: Week 52 (end of treatment)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Mirabegron + Solifenacin | Mirabegron + Propiverine | Mirabegron + Imidafenacin | Mirabegron + Tolterodine
Number analyzed (Participants) | 137 | 131 | 139 | 130
Participants | 26 | 21 | 21 | 14

16. Secondary Outcome: Change From Baseline in Postvoid Residual (PVR) Volume
Description: Measurement of PVR volume was made using either ultrasonography or urethral catheterization, provided that the same method was used for the same participant throughout the study.
Time Frame: Baseline and week 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: SAF
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Mirabegron + Solifenacin | Mirabegron + Propiverine | Mirabegron + Imidafenacin | Mirabegron + Tolterodine
Number analyzed (Participants) | 166 | 161 | 161 | 159
mL
  Week 4: number analyzed (Participants) | 162 | 157 | 158 | 157
  Week 4 | 9.07 (23.79) | 9.99 (36.05) | 6.81 (22.11) | 8.21 (28.58)
  Week 8: number analyzed (Participants) | 155 | 148 | 155 | 147
  Week 8 | 10.68 (34.38) | 3.23 (20.40) | 5.77 (25.39) | 8.39 (29.58)
  Week 12: number analyzed (Participants) | 144 | 146 | 145 | 142
  Week 12 | 4.72 (19.47) | 3.67 (20.42) | 7.19 (27.66) | 6.04 (28.98)
  Week 16: number analyzed (Participants) | 138 | 140 | 144 | 137
  Week 16 | 7.51 (22.06) | 1.06 (18.74) | 4.04 (20.69) | 8.67 (49.49)
  Week 20: number analyzed (Participants) | 133 | 138 | 141 | 134
  Week 20 | 2.32 (18.01) | 3.53 (19.43) | 2.97 (19.82) | 4.68 (27.56)
  Week 24: number analyzed (Participants) | 134 | 135 | 139 | 134
  Week 24 | 4.99 (21.14) | 4.03 (22.38) | 2.79 (16.06) | 1.46 (17.97)
  Week 28: number analyzed (Participants) | 133 | 133 | 140 | 133
  Week 28 | 2.95 (19.97) | 3.87 (19.82) | 5.56 (23.90) | 5.07 (29.92)
  Week 32: number analyzed (Participants) | 128 | 130 | 137 | 129
  Week 32 | 0.70 (16.90) | 1.34 (17.28) | 2.19 (17.26) | 3.11 (25.17)
  Week 36: number analyzed (Participants) | 128 | 130 | 137 | 129
  Week 36 | 4.11 (19.17) | 0.66 (17.96) | 2.18 (19.97) | 3.12 (17.85)
  Week 40: number analyzed (Participants) | 128 | 130 | 130 | 126
  Week 40 | 6.03 (21.79) | 3.29 (23.24) | 5.19 (23.09) | 5.40 (35.27)
  Week 44: number analyzed (Participants) | 128 | 128 | 128 | 123
  Week 44 | 2.17 (16.40) | 1.03 (16.89) | 3.14 (21.56) | 0.50 (18.59)
  Week 48: number analyzed (Participants) | 128 | 126 | 127 | 123
  Week 48 | 2.60 (16.30) | 0.71 (17.05) | 2.22 (17.58) | 2.33 (26.90)
  Week 52: number analyzed (Participants) | 127 | 128 | 125 | 123
  Week 52 | 3.56 (17.51) | 4.58 (22.19) | 2.84 (19.94) | 2.02 (24.67)
  End of treatment: number analyzed (Participants) | 164 | 160 | 161 | 159
  End of treatment | 8.17 (39.42) | 6.83 (32.20) | 4.52 (23.51) | 5.94 (35.83)

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to week 52
Description: Safety Analysis Set (SAF). The SAF consisted of participants who received at least 1 dose of the study drug for the treatment period.
Arm/Group | Mirabegron + Solifenacin | Mirabegron + Propiverine | Mirabegron + Imidafenacin | Mirabegron + Tolterodine
All-Cause Mortality (participants affected / at risk) | 0/166 | 0/161 | 0/161 | 1/159
Serious Adverse Events (participants affected / at risk) | 10/166 | 4/161 | 5/161 | 9/159
Other Adverse Events (participants affected / at risk) | 115/166 | 117/161 | 108/161 | 97/159
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mirabegron + Solifenacin (N=166) | Mirabegron + Propiverine (N=161) | Mirabegron + Imidafenacin (N=161) | Mirabegron + Tolterodine (N=159)
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 1 | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Disuse syndrome (General disorders) | 0 | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Chronic hepatitis C (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Vestibular neuronitis (Infections and infestations) | 0 | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Lung adenocarcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Spinal operation (Surgical and medical procedures) | 0 | 0 | 0 | 1
Cataract operation (Surgical and medical procedures) | 1 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
Microscopic polyangiitis (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mirabegron + Solifenacin (N=166) | Mirabegron + Propiverine (N=161) | Mirabegron + Imidafenacin (N=161) | Mirabegron + Tolterodine (N=159)
Tinnitus (Ear and labyrinth disorders) | 0 | 4 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 4
Cataract (Eye disorders) | 1 | 0 | 1 | 4
Abdominal discomfort (Gastrointestinal disorders) | 7 | 4 | 4 | 2
Constipation (Gastrointestinal disorders) | 37 | 27 | 24 | 19
Dental caries (Gastrointestinal disorders) | 0 | 6 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 4 | 2
Dry mouth (Gastrointestinal disorders) | 32 | 51 | 40 | 40
Dyspepsia (Gastrointestinal disorders) | 0 | 5 | 1 | 1
Gastritis (Gastrointestinal disorders) | 2 | 5 | 4 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 6 | 4 | 5
Vomiting (Gastrointestinal disorders) | 1 | 2 | 5 | 3
Malaise (General disorders) | 2 | 2 | 4 | 2
Cystitis (Infections and infestations) | 18 | 13 | 25 | 10
Gastroenteritis (Infections and infestations) | 3 | 2 | 5 | 2
Nasopharyngitis (Infections and infestations) | 35 | 39 | 34 | 32
Periodontitis (Infections and infestations) | 0 | 4 | 1 | 2
Pharyngitis (Infections and infestations) | 6 | 4 | 4 | 2
Oral herpes (Infections and infestations) | 4 | 2 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 4 | 6 | 3 | 5
Blood creatine phosphokinase increased (Investigations) | 1 | 1 | 4 | 3
Electrocardiogram QT prolonged (Investigations) | 1 | 2 | 5 | 1
Residual urine volume increased (Investigations) | 6 | 8 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 5 | 6 | 4
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 | 2 | 3 | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 5 | 2 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 1
Dizziness (Nervous system disorders) | 2 | 5 | 0 | 3
Headache (Nervous system disorders) | 5 | 4 | 0 | 2
Dysuria (Renal and urinary disorders) | 8 | 4 | 3 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 3 | 7 | 2 | 2
Eczema (Skin and subcutaneous tissue disorders) | 5 | 2 | 6 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi center data. Sponsor must receive a site's manuscript prior to publication for review and comment.